CLINICAL TRIAL: NCT00245349
Title: Biodistribution and Radiation Dosimetry of F-18 Fluorothymidine (FLT) Imaged With Positron Emission Tomography (PET) in Patients With Head and Neck Cancer: A Radioactive Drug Research Committee (RDRC) Study
Brief Title: Study to Calculate the Radiation Dosimetry in Subjects With Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: University of Iowa (Other)
Responsible Party: Yusuf Menda, M.D., University of Iowa Hospitals & Clinics
Other Study IDs: 200502799
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Last update posted 2008-06-10 (Estimated); Status verified 2008-06

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck cancer; Squamous cell carcinoma; FLT; Fluorothymidine; F-18
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor biopsy, blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- FLT: Study group receiving FLT for imaging
  Interventions: Procedure: F-18 Fluorothymidine

INTERVENTIONS:
Procedure: F-18 Fluorothymidine

SUMMARY:
Preliminary observations suggest positron emission tomography (PET) imaging with an F-18 labeled thymidine analog (FLT) can selectively identify proliferating and non-proliferating tissues, including tumors. FLT uptake in the tumor appears to reflect the level of cells undergoing DNA synthesis. This is clinically important because cell proliferation markers have significant prognostic value, both prior to initiating radiotherapy and as they change during the course of therapy. In the proposed study, the researchers assess the biodistribution and radiation dosimetry of FLT to obtain the necessary data to file an Investigational New Drug (IND) application with the Food and Drug Administration (FDA). The information collected under Radioactive Drug Research Committee (RDRC) approval will not be used for diagnostic purposes, to assess the subject's response to therapy, or for clinical management of the subject.

DETAILED DESCRIPTION:
There are approximately 40,000 new cases of head and neck cancer each year in the United States. Worldwide more than 500,000 individuals will develop head and neck cancer each year, ranking as the sixth most common cancer. These cancers are predominately squamous cell cancers. Approximately two thirds of subjects will present with locally advanced disease with either large disease at the primary site and/or spread to regional lymph node levels.

Despite aggressive treatment, 5-year survival remains poor (overall, approximately 50%). The major site of treatment failure is within the head and neck region, with distant metastases occurring in approximately 25% of subjects and usually after local and/or regional (nodal) failure.

Current treatment options for locally advanced head and neck cancer include combinations of surgery, radiation therapy, and chemotherapy. It is currently difficult to predict which combination will be best suited for any particular individual. Rapid methods of assessing the response of subjects to chemo-radiotherapy would be a useful tool, as it would permit the oncologist to change therapies, either in type or degree, in cases when the subject does not respond to the initial therapy regimen. Current best methods of evaluating tumor response are either serial CT examinations, so that changes in tumor size can be estimated or a fluorodeoxyglucose (FDG) positron emission tomography (PET) study in which changes in the metabolic status of the tumor are evaluated. Unfortunately, the anatomic information afforded by CT examinations often require months after treatment to allow the full effects of therapy to take place. Even after this time, the metabolic activity of any remaining tissue is nearly impossible to assess by CT scan, making it difficult to distinguish between fibrosis and viable tissue. Generally the FDG studies require 3-4 weeks after the end of the therapeutic regime before the relevant information is available, with more reliable information obtained at 3-4 months after treatment.

It is predictable that the most immediate signal of an anti-tumor therapeutic regime that has been successful is that the tumor cells will stop dividing (proliferating) after the therapy is initiated. Therefore, a tracer which is taken up into and retained in cells as a function of their proliferative activity should provide rapid information as to the effectiveness of the treatment. It is the objective of this study to determine the biodistribution and radiation dosimetry of tracer F-18 3'-deoxy-3'-fluorothymidine. This distribution data is essential before an Investigational New Drug (IND) application can be filed with the FDA that would allow the use of this tracer in clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to sign a written informed consent document.
2. Subject must have histologically confirmed stage III, or IV squamous cell carcinoma of the head and neck whose primary origin was from the oral cavity, oropharynx, hypopharynx, or larynx. Carcinoma must be staged using the American Joint Committee on Cancer (AJCC) staging criteria version 6. Adequate tumor must be amenable to biopsy via outpatient methods, therefore the majority of subjects will be those with oropharyngeal lesions.
3. Subjects must be scheduled to receive combined chemo-radiotherapy treatment for their standard cancer care. Treatment decisions will be made by the treating otolaryngologist, radiation, and medical oncologists.
4. Males or females greater than or equal to 21 years of age. Squamous cell cancer of the head and neck is exceedingly rare in children and not generally applicable to the pediatric population.
5. Karnofsky score greater than or equal to 60% at time of screening.
6. Life expectancy of greater than 6 months.
7. Subject must have normal organ and marrow function as defined below:

   * leukocytes greater than or equal to 3,000/microL
   * absolute neutrophil count greater than or equal to 1,500/microL
   * platelets greater than or equal to 100,000/microL
   * total bilirubin within normal institutional limits
   * AST(SGOT)/ALT(SGPT) less than or equal to 2.5 X institutional upper limit of normal
   * creatinine within normal institutional limits
   * BUN within normal institutional limits
   * PT and PTT < 2.0 X upper normal limits
8. The effects of FLT on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. A screening urine hCG will be administered to women of childbearing potential before each FLT scan.

Exclusion Criteria:

1. Subjects who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
2. Subject may not be receiving any other investigational agents.
3. Subject with a Karnofsky score below 60.
4. Pregnant women are excluded from this study. FLT PET has the potential for teratogenic effects. Because there are potentially unknown risks for adverse events in nursing infants secondary to treatment of the mother with FLT, breastfeeding should be discontinued if the mother is imaged with FLT and may not resume for 48 hours after the FLT imaging.
5. Subject with an inadequate marrow reserve as determined by history and/or the above tests.
6. Subject with a bleeding or clotting dysfunction as determined by medical history and above tests.
7. Subjects taking nucleoside analog medications such as those used as antiretroviral agents.
8. Inadequate tumor volume to allow for 2 biopsies.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Head & Neck Cancer
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2005-10; Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Menda, MD, Principal Investigator — University of Iowa, Department of Radiology-Nuclear Medicine; Kenneth J Dornfeld, MD, PhD, Principal Investigator — University of Iowa; Timothy Tewson, PhD, Principal Investigator — University of Iowa, Department of Radiology-Nuclear Medicine
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States